CLINICAL TRIAL: NCT05479071
Title: Relation of Antibodies Against Oxidized Low Density Lipoproteins to Disease Activit y and Cardiovascular Affection in Systemic Lupus.
Brief Title: Relation of Antibodies Against Oxidized Low Density Lipoproteins to Disease Activity and Cardiovascular Affection in Systemic Lupus.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, HADDEEL AHMED MOHMED SAYED AHMED, Dr, Assiut University
Other Study IDs: SLE
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: SLE
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SLE patients WITH cardiovascular disease: Relation of antibodies against LDL to disease activity in pt with cardiovascular disease
  Interventions: Diagnostic Test: Blood test
- SLE Patients without cardiovascular disease: Relation of antibodies against LDL to disease activity in pt without cardiovascular disease
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — Screening of antibodies against LDL

SUMMARY:
The aim of this study is to correlate the autoantibody against oxidized LDL with disease activity and cardiovascular affection in patients with SLE.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an autoimmune inflammatory disease affecting mainly women of fertile age. It is characterized by hyperactivity of B-cells and by overproduction of autoantibodies without organ specificity, many of which contribute to the formation of immunocomplexes. Their deposition in tissues and blood vessels results in inflammatory organ impairment (Khairy et al., 2017). As for the laboratory findings in SLE, production of autoantibodies without organ specificity aimed at nuclear, cytoplasmic, and surface antigens of the patient's body is typical. The most common SLE manifestations include involvement of skin, joints, cardiovascular system, lungs, renal glomeruli, central nervous system or hematopoiesis.

SLE can result in failure of the involved organs, severe forms of SLE thus bein gassociated with significant mortality (Pashnina et al., 2021).

Cardiovascular involvement is associated with increased morbidity and mortality of SLE patients. The most common SLE-related cardiovascular events are myocardial infarctions (MIs), cerebrovascular events, thromboembolic events (TEs), heart failure, and sudden death.

Cardiovascular events are proportionally higher in SLE compared to general populations of comparable age and sex (Ramirez et al., 2020). The pathogenic mechanisms of different cardiac diseases in SLE are still incompletely understood. Traditional risk factors for Cardiovascular affection, such as older age, high blood pressure (BP), high cholesterol and triglycerides, smoking, obesity, diabetes mellitus, and - last but not least - SLE therapy all play a critical role. These factors alone cannot adequately explain the increased incidence of cardiovascular disease commonly reported in patients with SLE. Metabolic syndrome was considered a remarkable risk factor for the development of subclinical atherosclerosis and increased carotid intima-media thickness The non-traditional biomarkers included both leptin and homocysteine, where leptin acts on the immune system as aproinflammatory cytokine. It promotes the proliferation and activation of T lymphocytes and induces production of Th1 cytokines. Homocysteinelevels have been identified as a predictor of atherosclerosis in patients with SLE, in whom high levels may be predictive levels of coronary calcification, platelet progression and increased IMT (Khairy et al., 2017).

Specific antibodies cause oxidation of low density lipoprotein (LDL) particles, thus accentuating their atherogenic effect, or exert a negative influence on the character of physiologically protective High density lipoprotein (HDL) particles. Endothelial dysfunction within the vascular system ensues, increasing its vulnerability, affinity to lipoproteins and activity of enzymes accelerating the development of atherosclerosis (Li et al., 2020).

LDLs are transported into artery walls, where they become trapped and bound in the extracellular matrix of the subendothelial space. These trapped LDLs are then seeded with reactive oxygen species produced by nearby artery wall cells, resulting in the formation of proinflammatory Oxidized LDL (OxLDL). oxLDL plays an important role in atherogenesisand may contribute to the immune activation and inflammation present in the atherosclerotic lesions, because it has chemotactic, immune-stimulatory, and toxic properties and is taken up by macrophages and other cells in the atherosclerotic plaque, which develop into foam cells. Epitopes characteristic of oxidized LDL can be found in atherosclerotic lesions by immunocytochemical techniques and atherosclerotic lesions contain immunoglobulins that recognize oxLDL (Ammar et al., 2021).

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients aged ≥ 18 years. 2. Patients fulfilling the American College of Rheumatology (ACE) criteria for SLE (Aringer et al., 2019).

3. Patients diagnosed with SLE and without cardiovascular disease (CVD) impairment before the diagnosis of SLE was established.

Exclusion Criteria:

1. Patients aged less than18 years.
2. Patients not fulfilling the American College of Rheumatology (ACE) criteria for SLE (Aringer et al., 2019).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients in our study will be subjected to:
  * History taking including: age, sex, special habit, BMI, comorbid diseases.
  * Pharmacological history.
  * Abdominal, neurological and locomotor systems examination.
  * Laboratory tests including:
    * Current activity of antibodies (antinucleolar antibodies (ANA)
      -, antinucleosomal antibodies, and anticardiolipin antibodies).
    * High sensitivity C-reactive protein (hsCRP)
    * oxidized LDL (oxLDL).
    * Lipid spectrum analysis comprised: the total cholesterol, LDL- cholesterol concentration, and HDL-cholesterol concentration.
  * ECG, and Echo.
  * Carotid intima- media thickness by carotid doppler.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Checking level of oxidized LDL. | Baseline
  We expect that oxidized LDL is increasing in patient with SLE and those patients will be at risk for cardiovascular disaeses.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu R, Svenungsson E, Gunnarsson I, Haegerstrand-Gillis C, Andersson B, Lundberg I, Elinder LS, Frostegard J. Antibodies to adult human endothelial cells cross-react with oxidized low-density lipoprotein and beta 2-glycoprotein I (beta 2-GPI) in systemic lupus erythematosus. Clin Exp Immunol. 1999 Mar;115(3):561-6. doi: 10.1046/j.1365-2249.1999.00830.x. PMID 10193434
- [Result] Wu R, Svenungsson E, Gunnarsson I, Andersson B, Lundberg I, Schafer Elinder L, Frostegard J. Antibodies against lysophosphatidylcholine and oxidized LDL in patients with SLE. Lupus. 1999;8(2):142-50. doi: 10.1191/096120399678847434. PMID 10192509
- [Result] Kurien BT, Scofield RH. Autoimmunity and oxidatively modified autoantigens. Autoimmun Rev. 2008 Jul;7(7):567-73. doi: 10.1016/j.autrev.2008.04.019. Epub 2008 May 27. PMID 18625446
- [Result] Tektonidou MG. Cardiovascular disease risk in antiphospholipid syndrome: Thrombo-inflammation and atherothrombosis. J Autoimmun. 2022 Apr;128:102813. doi: 10.1016/j.jaut.2022.102813. Epub 2022 Mar 2. PMID 35247655
- [Result] Tso TK, Huang WN. Elevation of fasting insulin and its association with cardiovascular disease risk in women with systemic lupus erythematosus. Rheumatol Int. 2009 May;29(7):735-42. doi: 10.1007/s00296-008-0781-7. Epub 2008 Nov 27. PMID 19037607